CLINICAL TRIAL: NCT03650140
Title: PKPD of Anthocyanins After Oral Cherry Juice Concentrate in Gout Patients
Brief Title: Pharmacokinetics and Pharmacodynamics of Anthocyanins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Naomi Schlesinger, MD, Professor of Medicine, Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro20170001180
Record Dates: First submitted 2018-08-13; First posted 2018-08-28 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Gout
Keywords: Gout; Tart Cherry; Pharmacokinetics
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tart cherry concentrate 60 mL (Active Comparator): Subjects will receive a single oral dose of 60 mL tart cherry concentrate. After a 2 week wash-out subjects will cross over into the 120 mL dose group.
  Interventions: Dietary Supplement: Tart cherry extract 60 mL; Dietary Supplement: Tart cherry extract 120 mL
- Tart cherry concentrate 120 mL (Active Comparator): Subjects will receive a single oral dose of 120 mL tart cherry concentrate. After a 2 week wash-out subjects will cross over into the 60 mL dose group.
  Interventions: Dietary Supplement: Tart cherry extract 60 mL; Dietary Supplement: Tart cherry extract 120 mL

INTERVENTIONS:
Dietary Supplement: Tart cherry extract 60 mL — Subjects will receive a single 60 mL oral dose of tart cherry extract.
Dietary Supplement: Tart cherry extract 120 mL — Subjects will receive a single 120 mL oral dose of tart cherry extract.

SUMMARY:
The purpose of the study is to establish the pharmacokinetic parameters of cherry juice concentrate and identify its potential to alter inflammatory markers in gout patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gout

Exclusion Criteria:

* Allergy to cherries or cherry products
* Any history of malignancy
* History of any pancreatic or biliary tract disease
* Significant Anemia
* History of significant renal (sCr > 1.5 mg/dL)
* Hepatic disease (liver enzymes 3 times upper limit of normal)
* Any active gastrointestinal condition
* History of large bowel resection for any reason
* Use of cherry juice concentrate or consumption of cherries within 14 days
* Personal or inherited bleeding disorders or currently on anticoagulation
* Women of childbearing age not on oral contraceptives
* Women who are pregnant or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Highly sensitive C-reactive protein (hs-CRP) | Maximal change in hs-CRP from baseline through study completion (during the 12 hours after a dose)
  Reduction in hs-CRP

SECONDARY OUTCOMES:
Area under the curve (AUC) | Through study completion (during the 12 hours after a dose)
  The area under the plasma anthocyanin concentration-time curve
Change in inflammatory marker expression | Through study completion (during the 12 hours after a dose)
  Fold change in mRNA expression of Nrf2
Peak plasma concentration (Cmax) | Through study completion (during the 12 hours after a dose)
  Peak plasma concentration of anthocyanins
Time to peak plasma concentration (Tmax) | Through study completion (during the 12 hours after a dose)
  Time to achieve peak plasma anthocyanin concentration
Half-life (t1/2) | Through study completion (during the 12 hours after a dose)
  Plasma anthocyanin half-life

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Schlesinger, MD, Principal Investigator — Robert Wood Johnson Medical School/ Rutgers RWJMS Gout Center
Locations (1):
- Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT03650140/ICF_000.pdf